CLINICAL TRIAL: NCT01119807
Title: Intraosseous Versus Intravenous Vascular Access During Cardiac Arrest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MeckIO2010
Record Dates: First submitted 2010-05-06; First posted 2010-05-10 (Estimated); Results first posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2021-11

CONDITIONS: Cardiac Arrest
Keywords: Intraosseous infusion; Emergency Medical Services
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intra Venous Access (Experimental): Patient initially receives IV access during resuscitation
  Interventions: Device: Intravenous access during OHCA
- Humeral IO (Experimental): Patient receives humeral IO access during resuscitation
  Interventions: Device: Humeral IO insertion
- Tibial IO (Active Comparator): Patient receives tibial IO access during resuscitation
  Interventions: Device: TIbial IO insertion

INTERVENTIONS:
Device: Intravenous access during OHCA — First attempt will be a peripheral IV in the AC. If this fails, second attempt will be a tibial IO, followed by a humeral IO when indicated.
  Arms: Intra Venous Access
Device: Humeral IO insertion — First attempt will be a humeral IO. Second attempt should occur at the tibia if the first humeral IO fails. Subsequent attempts will be for a peripheral IV or additional IOs as determined by the paramedic.
  Arms: Humeral IO
Device: TIbial IO insertion — First attempt will be a tibial IO. Second attempt should occur on the opposite tibia if the first IO fails. Subsequent attempts will be for a humeral IO or peripheral IV as selected by the paramedic.
  Arms: Tibial IO

SUMMARY:
The objective of this study will be to compare humeral and tibial IO needle insertions to peripheral IV access during cardiac arrest.

Hypothesis There is a difference in first attempt success of tibial IOs compared to humeral IOs or peripheral IV among cardiac arrest patients.

This was a randomized trial of adult patients experiencing a medical OOHCA where resuscitation efforts were initiated. Patients were randomized to 1 of 3 routes of vascular access. Prior to every shift, paramedics were distributed a randomly selected note card indicating the prescribed route for vascular access: tibial IO, humeral IO, or peripheral IV.

The selected method applied to the first attempt at vascular access only. Paramedics received intensive training and exposure to all three methods prior to study initiation. The primary outcome was first attempt success defined as secure needle position in the marrow cavity or a peripheral vein with normal fluid flow. Needle dislodgement during resuscitation was counted as a failure to maintain vascular access. In order to detect a statistical difference in the frequency of first attempt success a minimum of 50 patients for each arm of the study were needed.

DETAILED DESCRIPTION:
The objective of this study will be to compare humeral and tibial IO needle insertions to peripheral IV access during cardiac arrest.

Hypothesis There is a difference in first attempt success of tibial IOs compared to humeral IOs or peripheral IV among cardiac arrest patients.

Methods This will be a randomized controlled trial conducted within Mecklenburg County by the Mecklenburg County EMS Agency (MEDIC). The study population includes all adult (greater than 18 years of age) cardiac arrest patients of a medical etiology upon whom resuscitative efforts are initiated.

Patient Care Protocols Prehospital protocols for adult cardiac arrest patients within Mecklenburg County state that all first responders follow advanced cardiac life support (ACLS) algorithms during cardiopulmonary resuscitation. Current MEDIC protocols specify that initial vascular access be obtained by paramedics via either tibial or humeral IO needle insertion, followed by peripheral IV for secondary access. This study will randomize initial vascular access to a humeral IO, tibial IO, or peripheral IV.

Once paramedics arrive on-scene, they will take a pack from the ambulance containing all necessary supplies to begin resuscitation. These packs are already present on each ambulance in Mecklenburg County and contain an EZ-IO drill, IO needles, ACLS medications, and KING LTD airway device. For the purposes of this study, peripheral IV start kits will be added to these resuscitation packs at the start of study implementation.

Randomization Process

150 note cards will be prepared in advance and labeled with a vascular access method. [50 cards with "Tibial IO", 50 cards "Humeral IO", 50 cards with "Peripheral IV"] Each note card will be sealed in a blank, numbered envelope. A master list will be prepared in advance according to envelope number indicating which vascular access method was placed in each numbered envelope. This list will only be available to the MEDIC Quality Assurance/Quality Improvement (QA/QI) personnel responsible for paramedic debriefing and recirculation of unused envelopes.

Sealed envelopes will then be shuffled and placed at the MEDIC circulation window where resuscitation packs and ambulance equipment are distributed daily.

Each crew will randomly select and open an envelope prior to every shift. By opening the envelope at the start of the day, this will eliminate the possibility of envelopes being left in the ambulance unit or lost at the scene, as well as prevent delays with patient care.

The envelope number will be recorded at the circulation window indicating the specific MEDIC ambulance unit and assigned crew.

The vascular access route selected will apply to the crew's first cardiac arrest of the day.

Resuscitation Protocol

Paramedics will conduct the resuscitation according to existing procedure, and will proceed with vascular access as follows depending on the method selected by randomization:

Tibial IO First attempt will be a tibial IO. Second attempt should occur on the opposite tibia if the first IO fails. Subsequent attempts will be for a humeral IO or peripheral IV as selected by the paramedic.

Humeral IO First attempt will be a humeral IO. Second attempt should occur at the tibia if the first humeral IO fails. Subsequent attempts will be for a peripheral IV or additional IOs as determined by the paramedic.

Peripheral IV First attempt will be a peripheral IV in the AC. If this fails, second attempt will be a tibial IO, followed by a humeral IO when indicated.

Since it is extremely rare for any crew to conduct more than one cardiac arrest on a given day, the randomized vascular access method will only apply to the first cardiac arrest of the day. As crews do not return to the distribution center until the end of a shift (12 hours), it will be impossible to select additional envelopes for subsequent patient encounters. Paramedics will proceed with vascular access per current MEDIC prehospital protocols for any further cardiac arrest resuscitations that day.

If there is a contraindication to the vascular access site selected such as extremity amputations, orthopedic hardware, skin infection, or traumatic injuries, paramedics will proceed to the next insertion site as per the above protocol. For instance, if a patient with bilateral lower extremity amputations is randomized to a tibial IO insertion site, paramedics will classify this as a failed attempt and proceed to humeral IO, then peripheral IV as stated above. For patients with isolated skin infections or orthopedic hardware involving one extremity, paramedics will select the unaffected extremity for the first attempt. Any unforeseen circumstances will be addressed according to the paramedics' discretion and reported to the primary investigator immediately. Such occurrences will be included in the final data analysis for this study.

ELIGIBILITY:
Inclusion Criteria:

1. All cardiac arrests of a medical nature in patients greater than or equal to 18 years of age occuring in Mecklenburg county, NC.

Exclusion Criteria:

1. Traumatic cardiac arrests - different prehospital protocols exist for resuscitations involving traumatic arrests (i.e. motor vehicle accidents, motorcycle accidents, falls, and penetrating injuries including stabbings and gunshot wounds).
2. Cardiac arrests due to hemorrhage - for the purposes of this study, such arrests are not considered to be of a "medical etiology" since massive blood loss is the contributing factor and only rapid volume resuscitation is indicated.
3. Cardiac arrests involving children or young adults - any patient less than 18 years of age will be excluded as different prehospital protocols exist for children in cardiac arrest. Age verification will occur upon data collection using patient date of birth when available. Any data collected from a patient found to be less than 18 years of age after resuscitation, will also be excluded from data analysis.
4. Patients with established vascular access prior to cardiac arrest - patients who deteriorate during transport into cardiac arrest but already have a peripheral IV or IO needle established will be excluded from the study. Randomization cannot be applied to these encounters as vascular access has already been selected and documentation by a sole provider is not possible during transport.
5. Patients with a Do Not Resuscitate (DNR) - in some circumstances, cardiopulmonary resuscitation is initially performed on patients until a DNR order is produced. These patients will be excluded from the study as the full protocol cannot be implemented.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2010-05; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Studnek, PhD, Study Director — Mecklenburg EMS Agency
Locations (1):
- Mecklenburg EMS Agency, Charlotte, North Carolina, United States

REFERENCES:
- [Result] Reades R, Studnek JR, Vandeventer S, Garrett J. Intraosseous versus intravenous vascular access during out-of-hospital cardiac arrest: a randomized controlled trial. Ann Emerg Med. 2011 Dec;58(6):509-16. doi: 10.1016/j.annemergmed.2011.07.020. PMID 21856044

RESULTS

PARTICIPANT FLOW:
Groups:
- Intravenous: Intravenous access during OHCA: First attempt will be a peripheral IV in the AC. If this fails, second attempt will be a tibial IO, followed by a humeral IO when indicated.
Period: Overall Study
Arm/Group | Intravenous | Humeral IO | Tibial IO
Started | 67 | 51 | 64
Completed | 67 | 51 | 64
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous | Humeral IO | Tibial IO | Total
Number analyzed (Participants) | 67 | 51 | 64 | 182
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (2) | 61 (2) | 66 (2) | 64 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 15 | 23 | 80
  Male | 25 | 36 | 41 | 102
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 32 | 21 | 35 | 88
  Race: Other | 35 | 30 | 29 | 94
Region of Enrollment [Number; unit: participants]
  United States | 67 | 51 | 64 | 182

OUTCOME MEASURES:

1. Primary Outcome: First Attempt Success Rate Between the Tibial IO, Humeral IO, and Peripheral IV.
Description: This measure will be assessed on the day an individual experiences cardiac arrest and will not be followed upon admission to the emergency department.
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous | Humeral IO | Tibial IO
Number analyzed (Participants) | 67 | 51 | 64
Participants | 26 | 17 | 58

ADVERSE EVENTS:
Arm/Group | Intravenous | Humeral IO | Tibial IO
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/51 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/51 | 0/64
Other Adverse Events (participants affected / at risk) | 0/67 | 0/51 | 0/64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No